CLINICAL TRIAL: NCT07208643
Title: Long-term Stability of Peri-implantitis Treatments: a 3-year Clinical Evaluation
Status: Not yet recruiting | Type: Observational
Sponsor: Ramón Pons Calabuig (Other)
Responsible Party: Sponsor-Investigator, Ramón Pons Calabuig, dds ms, Universitat Internacional de Catalunya
Organization: Universitat Internacional de Catalunya (Other)
Other Study IDs: PER-ECL-2025-03; PER-ECL-2025-03 (Registry Identifier: CEIm de la Clínica Universitària d'Odontologia de la UIC); Long-term stability of peri-im (Other: CEIm de la Clínica Universitària d'Odontologia de la UIC)
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Peri-implantitis
Keywords: Peri-implantitis; Non-surgical therapy; Reconstructive therapy; Maintenance therapy; Prospective study; flapless treatment
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 'atients previously enrolled in the PER-ECL-2019-05 trial: Initially, 36 patients with advanced peri-implantitis were enrolled in a randomized clinical trial evaluating the clinical, radiographic and patient-related outcomes of reconstructive therapy following a non-surgical phase of peri-implantitis treatment compared to non-surgical treatment alone (PER-ECL-2019-05) .At the study conclusion 34 patients were re-evaluated and 2 patients were excluded from the study

SUMMARY:
This prospective study will include patients previously enrolled in the PER-ECL-2019-05 trial who attend the Department of Periodontology (CUO) for maintenance therapy or treatment of periodontal and/or peri-implant diseases, provided they meet the inclusion criteria.

Initially, 36 patients with advanced peri-implantitis were enrolled in a randomized clinical trial evaluating the clinical, radiographic and patient-related outcomes of reconstructive therapy following a non-surgical phase of peri-implantitis treatment compared to non-surgical treatment alone (PER-ECL-2019-05) (10).

At the study conclusion 34 patients were re-evaluated and 2 patients were excluded from the study (10).

In the original study, adult patients presenting at least one titanium implant diagnosed with peri-implantitis were identified among patients referred to the Department of Periodontology of UIC between January 2020 and October 2022. Peri-implantitis was diagnosed following the case definition of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions (11) that is, PPD ≥ 6 mm combined with bleeding on probing (BOP) and/or suppuration (SUP), together with progressive bone loss in relation to the radiographic bone level assessment. In those cases where initial radiograph was unavailable, the definition of a peri-implantitis case was based on radiographic evidence of bone level ≥3 mm apical to the most coronal portion of the intra-osseous part of the implant (12).

At the outset of the original study, participants were randomly assigned to one of two groups:

The first group received only non-surgical therapy for peri-implantitis, while the second group underwent a non-surgical phase followed by reconstructive surgical treatment. This design allowed for direct comparison of the clinical, radiographic, and patient-centered outcomes between the two treatment modalities. Both groups were managed and evaluated according to standardized protocols, ensuring consistency and reliability of the results at 12 months .

Patients who have not returned to the Department will be contacted by telephone and invited to participate through the academic office.

At 36 months, a single follow-up will be carried out including:

A detailed clinical examination. A standardized radiographic assessment.

DETAILED DESCRIPTION:
1. Introduction:

   There is a notable lack of comprehensive data regarding the long-term outcomes of surgical and non-surgical interventions for peri-implantitis. Most existing evidence stems from studies with 1 year follow-up or retrospective studies (1-5).

   The factors influencing the long-term stability of surgical treatment for peri-implantitis remain poorly understood. In a 7-year follow-up, Roccuzzo et al. (2017) observed that 50% of treated implants experienced recurrence of peri-implantitis, with retreatment needs being associated with implant surface characteristics (6). Similarly, Carcuac et al. (2020) found that 44% of implants showed disease recurrence after 5 years (7). More recently, Romandini et al. (2023) reported that approximately 20% of surgically treated implants were lost over a 4-year period, with implant failure being linked to the presence of baseline suppuration and the use of modified implant surfaces (4). Other studies, however, noted lower rates of recurrence/progression ranging from 20% to 32% during 3-5 years of follow-up (8,9).

   Conversely, evidence regarding the long-term outcomes of non-surgical treatment for peri-implantitis remains particularly scarce in the current literature, and to date, no studies have thoroughly investigated the factors associated with the stability of such therapeutic approaches.

   As part of a randomized controlled clinical trial evaluating the potential benefits of adjunctive reconstructive therapy in the management of advanced peri-implantitis, 36 patients were enrolled and followed for one year (10 ). The results indicated that both treatment strategies were moderately effective in achieving disease resolution. However, deeper baseline probing pocket depths were negatively associated with successful outcomes. Notably, sites treated with reconstructive surgical therapy demonstrated significantly greater marginal bone level gain. Despite this, the influence of improved bone support on the long-term maintenance of peri-implant health remains unclear. The present prospective study aims to elucidate further the factors associated with the long-term stability of both non-surgical and reconstructive treatment outcomes.
2. Objectives:

   This prospective study aims to evaluate the factors associated with the stability of the disease following non-surgical or reconstructive therapy.
3. Hypothesis:

   The non-surgical mechanical and antibiotic therapy of peri-implantitis in the treatment of infraosseous defects around implants will achieve similar stability at 36 months when compared to the same protocol and the adjunction of a regenerative surgical therapy by means of xenograft plus a collagen membrane.
4. Material and methods:

4.1 Study design: This document refers to the continuation of the original clinical study registered under protocol number PER-ECL-2019-05. The initial 1-year randomized controlled trial has been successfully completed, with all clinical and radiographic outcomes recorded and analyzed (10). Given the clinical importance of evaluating long-term stability in peri-implantitis treatment, the follow-up period has been extended to a total of 3 years. All participants who completed the 36-month study will be invited to take part in this extended observation phase, during which clinical and radiographic evaluations will be conducted at 36 months. This is a prospective clinical trial with 3-year follow-up.

4.2 Setting of the study: Patients previously enrolled in the study PER-ECL-2019-05 and attending the Department of Periodontology (CUO) for maintenance therapy or treatment of periodontal and/or peri-implant diseases will be included in the study. Patients who have not attended the Department of Periodontology (CUO) will be contacted by phone and invited to participate in the study by the academic secretary.

4.3 Study population: Initially, 36 patients with advanced peri-implantitis were enrolled in a randomized clinical trial evaluating the clinical, radiographic and patient-related outcomes of reconstructive therapy following a non-surgical phase of peri-implantitis treatment compared to non-surgical treatment alone (PER-ECL-2019-05) (10).

At the study conclusion 34 patients were re-evaluated and 2 patients were excluded from the study (10).

In the original study, adult patients presenting at least one titanium implant diagnosed with peri-implantitis were identified among patients referred to the Department of Periodontology of UIC between January 2020 and October 2022. Peri-implantitis was diagnosed following the case definition of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions (11) that is, PPD ≥ 6 mm combined with bleeding on probing (BOP) and/or suppuration (SUP), together with progressive bone loss in relation to the radiographic bone level assessment. In those cases where initial radiograph was unavailable, the definition of a peri-implantitis case was based on radiographic evidence of bone level ≥3 mm apical to the most coronal portion of the intra-osseous part of the implant (12).

At the outset of the study, participants were randomly assigned to one of two groups:

The first group received only non-surgical therapy for peri-implantitis, while the second group underwent a non-surgical phase followed by reconstructive surgical treatment. This design allowed for direct comparison of the clinical, radiographic, and patient-centered outcomes between the two treatment modalities. Both groups were managed and evaluated according to standardized protocols, ensuring consistency and reliability of the results at 12 months .

4.4. Inclusion/Exclusion criteria

Inclusion criteria:

1. Patiens previously enrolled in the randomized clinical trial PER-ECL-2019-05, which included 36 patients with advanced peri-implantitis.
2. Completion of the original study protocol, including either reconstructive surgical therapy following a non-surgical phase or non-surgical therapy alone.
3. Signed informed consent for participation in the follow-up assessment.

Exclusion criteria:

1. Did not complete the original clinical trial protocol (PER-ECL-2019-05) or withdrew before final evaluation.
2. Had the implant removed due to complications unrelated to peri-implantitis progression.
3. Have developed systemic diseases or conditions (e.g., uncontrolled diabetes, immunosuppression, malignancy) that may affect periodontal or peri-implant tissue healing or confound clinical outcomes.
4. Are currently undergoing antibiotic or antiresorptive therapy (e.g., bisphosphonates) that could interfere with bone metabolism.
5. Are pregnant or breastfeeding at the time of the follow-up visit.
6. Are unwilling or unable to attend the clinical follow-up appointment or provide informed consent.

4.5 Study visit

The single examination at 36 months will include:

4.5.1 Clinical examination Information regarding changes in medical history, and medication will be obtained. Smoking habit will be re- assessed [current smoker, former smoker, or never-smoker (12) and reported smoking exposure [pack-years: number of cigarettes smoked per day multiplied by the number of years the patient has smoked and divided by 20 (a standard pack of cigarettes)] (13) will be also registered.

Additionally, implant position and implant system will be recorded, as was the type of prosthesis (i.e., cemented/screw-retained).

All clinical examinations will be performed by a calibrated examiner (M.I.A.) using a UNC-15 periodontal probe. The intra-rater reliability for key implant-related variables (mesial PPD, BOP and plaque) will be assessed on the same day in 12 patients with 12 implants. The intra-class correlation coefficient (ICC) will be used to calculate the intra-rater reliability of continuous variables, while Cohen's Kappa (κ) will be used to assess the intra-rater reliability of categorical variables.

The clinical examination will include the assessments of the following variables (14):

1. Plaque index (PI), assessed as the presence or absence of plaque along the mucosal margin (15).
2. Bleeding on probing (BOP), dichotomously evaluated as the presence or absence of bleeding within 30 s after probing (16).
3. Suppuration on probing (SOP), dichotomously evaluated as the presence or absence of suppuration within 30 s after probing (16).
4. Peri-implant probing depth (PPD), calculated as the distance (mm) from the mucosal margin to the bottom of the peri-implant pocket (16).
5. Recession (REC), measured as the distance (mm) from the mucosal margin to the most apical portion of the crown (3).
6. Keratinized mucosa width (KMW), measured as the distance (mm) from the mucosal margin to the mucogingival junction.

In addition, the full-mouth plaque score (FMPS) will be calculated at the patient level by assigning a binary score to each surface (presence/absence of plaque) and calculating the percentage of total tooth/implant surfaces that revealed the presence of plaque detected by a periodontal probe (17).

4.5.2 Radiographic examination Radiographic examinations will be conducted at the same time points as described for the clinical assessments.

All peri-apical radiographs will be taken with an intra-oral phosphor plate using a long-cone parallel technique. Additionally, radiographs will be captured with the aid of an individualized silicone bite block (18) to ensure standardization and reproducibility of radiographic images. Radiographic measurements will be performed using image analysis software (ImageJ64; National Institutes of Health, Bethesda, MD, USA) by one previously calibrated examiner (R.P.). Calibration will be achieved by calculating the ICC after analyzing radiographic MBL on two separate occasions, 1 week apart. Radiographs will be calibrated in the image analysis software using the known implant dimensions as reference values. The following variables will be assessed on the radiographs:

* Mean bone level (MBL). The mean distance (mm) between the implant shoulder and the first visible bone-to-implant contact will be assessed at the mesial and distal aspects of each implant and the mean of the two values will be determined (1).
* Intrabony defect angle (AW). The angle resulting from a vertical line along the outer implant surface and a line extending along the peri-implant bone defect (1).

4.6 Outcomes: The primary outcome was recurrence/progression of peri-implantitis between years 1 and 3, defined as any of the following events: (a) bone loss >1.0 mm, (b) surgical retreatment, (c) implant removal/loss ) (7).

Secondary outcomes included changes (i.e., from baseline to 12 months) in (i) PPD, (ii) deepestPPD (PPDd), (iii) BOP, (iv) SOP, (v) plaque, (vi) buccal REC, (vii) buccal KMW, and (viii) MBL,evaluated at different time points. PPD was defined as the mean value of PPD measured at six sitesper implant, while PPDd referred to the deepest pocket recorded for each implant. Threshold values for PPD, BOP, SOP, plaque, buccal REC, MBL were also assessed at the 36-month follow-up.

5.Hypothesis:

4.4 Alternative hypothesis There is a significant difference in the recurrence or progression of peri-implantitis between treatment groups from year 1 to year 3, as measured by the incidence of bone loss >1.0 mm, surgical retreatment, or implant removal/loss.

6. Withdrawal of consent The Patient Information Sheet will clearly state that the patient can withdraw from the study at any time without prejudice or explanation.

7. Statistical analysis: The patient will be considered the unit of analysis. In order to describe the qualitative variables, absolute frequencies and percentages will be used. The description of quantitative variables will be performed using the mean, standard deviation (SD), median and quartiles. The Kolmogorov-Smirnov test will be used to assess the normality of distributions. An analysis will be carried out to determine differences in study outcomes between groups. Analysis will be based on the ITT (intention to treat) population using the last observation carried forward (LOCF) approach. The relationship between two qualitative variables will be calculated using the chi-squared test or Fisher's exact test (if in a given case the frequency observed is < 5). For ordinal variables, linear regression will be calculated using Kendall's tau coefficient.

Quantitative variables will be compared using the Student's t-test (< 2 categories), analysis of variance [ANOVA] (for variables > 2 categories), linear regression test and Scheffé's multiple comparisons test or U Mann Whitney non-parametric test. The linear relationship between the quantitative variables will be calculated using Pearson's correlation coefficient or Spearman's rank correlation test (if the variable is not normally distributed). Changes vs. baseline will be analyzed using the Wilcoxon non-parametric test or Mc Nemar test.

A final model will be developed using back stepwise logistic regression analysis including progression of peri-implantitis as a dependent variable. Variables with a significance of <0.2 in the univariate analysis will be included as independent variables. The results will be described with odds ratios (OR) with a 95% confidence interval (CI) and p-values.

Level of significance will be set at 0.05. The SPSS version 23.00 software (SPSS Inc., Chicago, IL, USA) will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patiens previously enrolled in the randomized clinical trial PER-ECL-2019-05, which included 36 patients with advanced peri-implantitis.

  2. Completion of the original study protocol, including either reconstructive surgical therapy following a non-surgical phase or non-surgical therapy alone.

  3.Signed informed consent for participation in the follow-up assessment.

Exclusion Criteria:

* 1.Did not complete the original clinical trial protocol (PER-ECL-2019-05) or withdrew before final evaluation.

  2.Had the implant removed due to complications unrelated to peri-implantitis progression.

  3.Have developed systemic diseases or conditions (e.g., uncontrolled diabetes, immunosuppression, malignancy) that may affect periodontal or peri-implant tissue healing or confound clinical outcomes.

  4.Are currently undergoing antibiotic or antiresorptive therapy (e.g., bisphosphonates) that could interfere with bone metabolism.

  5.Are pregnant or breastfeeding at the time of the follow-up visit. 6.Are unwilling or unable to attend the clinical follow-up appointment or provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patiens previously enrolled in the randomized clinical trial PER-ECL-2019-05, which included 36 patients with advanced peri-implantitis and treated with non surgical therapy or surgical therapy + reconstructive therapy
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
ecurrence/progression of peri-implantitis | 3 years
  The primary outcome was recurrence/progression of peri-implantitis between years 1 and 3, defined as any of the following events: (a) bone loss >1.0 mm, (b) surgical retreatment, (c) implant removal/loss )
recurrence/progression of peri-implantitis | 3 years
  The primary outcome was recurrence/progression of peri-implantitis between years 1 and 3, defined as any of the following events: (a) bone loss >1.0 mm, (b) surgical retreatment, (c) implant removal/loss )

CONTACTS AND LOCATIONS:
Overall Officials: CRISTINA VALLES CS VALLES, PhD, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Bacelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Soldini MC, Pons R, Nart J, Monje A, Carrio N, Valles C. Reconstructive Therapy of Peri-Implantitis Following Non-Surgical Treatment: A Randomized Controlled Trial. Clin Implant Dent Relat Res. 2025 Apr;27(2):e70024. doi: 10.1111/cid.70024. PMID 40183214